CLINICAL TRIAL: NCT00300391
Title: ORIC-I: Optimizing Recovery From Intensive Care: Mechanical Ventilation and Delirium
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment to meet aims.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Barb Early, MACRO Clinical Director, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0505051; 1K23HL078760-01A1 (NIH)
Record Dates: First submitted 2006-03-06; First posted 2006-03-08 (Estimated); Results first posted 2017-12-20 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-11

CONDITIONS: Delirium
Keywords: Delirium; Mechanical ventilation; Intensive care; Haloperidol
MeSH Terms: conditions — Delirium | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- haloperidol (Experimental): Once diagnosed as delirious, randomized to haloperidol 5 mg IV
  Interventions: Drug: haloperidol
- placebo (Placebo Comparator): once diagnosed as delirious, received 5 mg saline placebo
  Interventions: Other: Saline placebo

INTERVENTIONS:
Drug: haloperidol — Aim #1. To conduct a RCT of IV haloperidol vs. placebo for the treatment of delirium in mechanically ventilated ICU patients. Patients in the cohort study that go on to develop delirium will be enrolled in a RCT comparing treatment with scheduled haloperidol vs. placebo. By comparing differences between treatment and placebo groups, we will test the hypothesis that treatment with scheduled haloperidol improves the primary outcome of 28-day and 90 day mortality and secondary outcomes of total delirium days, duration of mechanical ventilation, and ICU length of stay.
  Other Names: Haldol
  Arms: haloperidol
Other: Saline placebo — control arem
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if treating delirious intensive care unit patients with haloperidol improves mortality.

DETAILED DESCRIPTION:
Intensive care unit delirium is a serious medical condition that is associated with increased morbidity and mortality. In this study, 304 delirious mechanically ventilated subjects will be randomized to haloperidol 5mg IV every 12 hours or placebo to determine if treatment with haloperidol improves short and long-term mortality.

ELIGIBILITY:
Inclusion Criteria:

* All adult (>=18 years of age) mechanically ventilated patients admitted to the medical, surgical, trauma, or cardiothoracic ICUs of the UPMC main campus who are expected by the ICU clinical team to require >24 hours of mechanical ventilation

Exclusion Criteria:

* Baseline QTc >480 milliseconds (ms); history of Parkinson's disease; pregnancy; history of schizophrenia or neurologic disease that would confound the delirium assessment; deafness or inability to understand English or Spanish; extubation prior to enrollment; previously enrolled in this study; patient, family, or attending physician refusal; death before enrollment; treatment with haloperidol within 2 days prior to ICU admission; and prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric B Milbrandt, MD, MPH, Principal Investigator — University of Pittsburgh Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milbrandt EB, Kersten A, Kong L, Weissfeld LA, Clermont G, Fink MP, Angus DC. Haloperidol use is associated with lower hospital mortality in mechanically ventilated patients. Crit Care Med. 2005 Jan;33(1):226-9; discussion 263-5. doi: 10.1097/01.ccm.0000150743.16005.9a. PMID 15644675

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was pre-maturely terminated and although sincere efforts were made to locate the relevant (and accurate) data for results reporting, limited data could be obtained and are reported in the Results section. Some data were either missing or were conflicting and were therefore, excluded.
Pre-assignment Details: 7 of 40 enrolled subjects never developed delirium, while 2 of 40 had persistent coma and died without ever opening eyes. Subjects were randomized to groups once the delirium was diagnosed. 31 subjects developed delirium and were eligible to randomized. 1 withdrew before starting/being randomized, as a result, 30 subjects were randomized.
Groups:
- Haloperidol: Once delirium was diagnosed, subjects were randomized to haloperidol 5 mg IV q 12h, which was continued until liberation from mechanical ventilation or 28 days, whichever was first.
- Placebo: Once delirium was diagnosed, subjects were randomized to identical placebo, which was continued until liberation from mechanical ventilation or 28 days, whichever was first.
Period: Overall Study
Arm/Group | Haloperidol | Placebo
Started | 16 | 14
Completed | 16 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haloperidol | Placebo | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Customized [Count of Participants; unit: Participants]
  >=18 Years | 16 | 14 | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: 28-day All-cause Mortality
Time Frame: Daily
Population: This study was pre-maturely terminated and although sincere efforts were made to locate the relevant and accurate data for results reporting, limited data could be obtained. Data are not available per-Arm (Haloperidol vs Placebo) for this Outcome Measure. The only available data are grouped by the "Delirium," "Persistent Coma," and "No delirium".
Measure: Count of Participants; unit: Participants
Groups:
- Delirium: Once diagnosed as delirious, randomized to haloperidol 5 mg IV
  haloperidol: Aim #1. To conduct a RCT of IV haloperidol vs. placebo for the treatment of delirium in mechanically ventilated ICU patients. Patients in the cohort study that go on to develop delirium will be enrolled in a RCT comparing treatment with scheduled haloperidol vs. placebo. By comparing differences between treatment and placebo groups, we will test the hypothesis that treatment with scheduled haloperidol improves the primary outcome of 28-day and 90 day mortality and secondary outcomes of total delirium days, duration of mechanical ventilation, and ICU length of stay.
Arm/Group | Delirium | Persistent Coma | No Delirium
Number analyzed (Participants) | 30 | 2 | 7
Participants | 4 | 2 | 1

2. Primary Outcome: 90-day All-cause Mortality
Time Frame: 90 Days from enrollment in study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Delirium | Persistent Coma | No Delirium
Number analyzed (Participants) | 30 | 2 | 7
Participants | 4 | 2 | 1

3. Secondary Outcome: Duration of Mechanical Ventilation
Time Frame: daily
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Delirium | Persistent Coma | No Delirium
Number analyzed (Participants) | 30 | 2 | 7
day | 4.5 [3 to 10] | 6 [4 to 8] | 4 [2 to 13]

4. Secondary Outcome: ICU Length of Stay
Time Frame: Daily
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | Delirium | Persistent Coma | No Delirium
Number analyzed (Participants) | 30 | 2 | 7
day | 9 [5 to 14] | 6 [4 to 8] | 7 [6 to 16]

ADVERSE EVENTS:
Time Frame: Limited data can be obtained to make sure AE data time frame. However, once the patient has left the ICU, data will no longer collect on a daily basis. On or about day 28 after enrollment and 90-days after enrollment, a research coordinator will contact the patient. For this 28-day and 90-day follow-up, the following were recorded 1) whether the patient is in the hospital and if not, where the patient was discharged to, and 2) if the patient is alive and if not, what the cause of death was.
Description: All the AEs were reported as the relationship to study drug. The following four cases were reported as very likely related to study drug. AEs were not reported as "Serious" or not in the limited data we found. All the AEs were listed in one table, and only Elevated QTc 494, 505, 548, 520 are very likely related to study drug, and the others are not related to study drug.
Arm/Group | Haloperidol | Placebo
All-Cause Mortality (participants affected / at risk) | 1/16 | 2/13
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/13
Other Adverse Events (participants affected / at risk) | 16/16 | 12/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haloperidol (N=16) | Placebo (N=13)
Elevated QTc .494 (Cardiac disorders) | 1 (1) | 0 (0)
Elevated QTc .505 (Cardiac disorders) | 1 (1) | 0 (0)
Elevated QTc 548 (Cardiac disorders) | 1 (1) | 0 (0)
Elevated QTc 520 (Cardiac disorders) | 0 (0) | 1 (1)
Hypoxemic resp failure ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Nosocomial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
RUL collapse (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bilateral infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Trachestomy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Abdominal surgery (closure) (Surgical and medical procedures) | 0 (0) | 1 (1)
Intrapulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachycardia, restlessness desat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OR-cleansing and closure of leg wound (Surgical and medical procedures) | 1 (1) | 0 (0)
Lower lobectomy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Self extubation with continued resp. insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
GU hemorrhage related to selfremoval of Foley catheter (Gastrointestinal disorders) | 1 (1) | 0 (0)
Reintubated for resp. insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Failure to wean from ventilator (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pseudomonas pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
MRSA (Infections and infestations) | 1 (1) | 1 (1)
ARF (Renal and urinary disorders) | 1 (1) | 0 (0)
VTach (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Viral pneumonia, ARDS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower extremity DVT (Vascular disorders) | 0 (0) | 1 (1)
Nosocomial pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation/delirium (Psychiatric disorders) | 4 (4) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
A Fib (Cardiac disorders) | 1 (1) | 0 (0)
Apnea/desaturation during weaning (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sedation interruption associated with desaturation and tachycardia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Failure to wean from ventilator (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Azotemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic hyponatremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastric and duodenal ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
Polymicrobial bilateral pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Hepatobiliary disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Lower GI bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Bacterial peritononitis (Infections and infestations) | 0 (0) | 1 (1)
ARD'S (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Extremity ischemia (Vascular disorders) | 1 (1) | 0 (0)
Acute renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
IVC (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
VATS/Empyema (Surgical and medical procedures) | 0 (0) | 1 (1)
Sacral decubitus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DVT (Vascular disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was pre-maturely terminated. Although sincere efforts were made to locate the relevant and accurate data, limited data could be obtained. Also, conflicting information was available with respect to participant enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No